CLINICAL TRIAL: NCT05352074
Title: STOPS Trial: A Multicentre Prospective Randomised Clinical Trial Comparing Total Colectomy With Ileorectal Anastomosis Versus Subtotal Colectomy With Cecal-rectal Anastomosis for Slow Transit Constipation
Brief Title: STOPS Trial: Total vs Subtotal Colectomy for Slow Transit Constipation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Weidong Tong, Director, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20211114
Record Dates: First submitted 2022-04-03; First posted 2022-04-28 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Slow Transit Constipation; Surgery
Keywords: Slow Transit Constipation; Total Colectomy with Ileorectal Anastomosis; Subtotal Colectomy with Caecorectal Anastomosis; Defecation Function; Quality of Life; Randomized Controlled Trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total colectomy with ileorectal anastomosis (Active Comparator): Total colectomy with ileorectal anastomosis (TC-IRA) serves as the standard surgical treatment for slow transit constipation.
  Interventions: Procedure: Total colectomy with ileorectal anastomosis
- Subtotal colectomy with cecal-rectal anastomosis (Experimental): Subtotal colectomy with cecorectal anastomosis (SC-CRA) is selectively employed for slow transit constipation.
  Interventions: Procedure: Subtotal colectomy with cecal-rectal anastomosis

INTERVENTIONS:
Procedure: Total colectomy with ileorectal anastomosis — Following complete colonic mobilization without preservation of the ileocolic vascular pedicle, the surgical specimen was extracted by extending the right lower quadrant trocar incision to approximately 4-5 cm. A resection of ileum, 2-3 cm proximal to the ileocecal junction, will be conducted by stapler. The anvil of a 29-mm circular stapler was inserted into the proximal ileal lumen and repositioned intra-abdominally. Ileorectal anastomosis was performed by transanal insertion of the circular stapler, aiming to achieve a tension-free, contamination-minimized reconstruction. Finally, a closed suction drain was placed in the rectouterine pouch (Douglas pouch), and all abdominal incisions were closed in layers.
  Arms: Total colectomy with ileorectal anastomosis
Procedure: Subtotal colectomy with cecal-rectal anastomosis — Following complete colonic mobilization with preservation of the ileocolic vascular pedicle and its branches, the surgical specimen was extracted by extending the right lower quadrant trocar incision to 4-5 cm. After insertion of the anvil from a 29-mm circular stapler through the ascending colon resection margin, a resection about 3 cm distal to the ileocecal junction will be conducted. The cecum was then positioned in the pelvis without rotational torsion, and an antiperistaltic cecorectal anastomosis was created between cecal fundus (after appendectomy) and the rectal stump. The anastomosis was performed via transanal insertion of the circular stapler to ensure tension-free, contamination-controlled reconstruction. Finally, a closed suction drain was placed in the rectouterine pouch (Douglas pouch), and all abdominal incisions were closed in a layered fashion.
  Arms: Subtotal colectomy with cecal-rectal anastomosis

SUMMARY:
Total colectomy with ileorectal anastomosis is a traditional surgical option for slow transit constipation (STC). Subtotal colectomy with caecorectal anastomosis have been reported to be a potential alternative approach. Thus, the optimal surgical option for STC is controversial.

DETAILED DESCRIPTION:
Constipation, a prevalent gastrointestinal disorder, affects 10%-15% of adults in the United States and approximately 8.2% of China's general population. Slow transit constipation (STC), accounting for 15%-42% of constipation cases, is characterized by impaired colonic motility. For patients refractory to conservative therapies who experience chronic, intractable symptoms and diminished quality of life (QoL), surgical intervention becomes the last-resort treatment. The primary surgical approach for STC has historically been total colectomy with ileorectal anastomosis (TC-IRA). Over the past two decades, however, subtotal colectomy with cecorectal anastomosis (SC-CRA) has garnered growing interest within the surgical community due to its potential to mitigate postoperative diarrhea. Despite this benefit, SC-CRA raises concerns about an elevated risk of recurrent constipation. The debate regarding the superiority of these approaches remains unresolved. This study aims to address this controversy through a comparative analysis of TC-IRA and SC-CRA, evaluating their therapeutic efficacy and safety profiles in refractory STC.

ELIGIBILITY:
Inclusion criteria

1. Patients (≥18 years of age) of either sex
2. Patients with conditions in agreement with the Roman IV criteria of functional constipation
3. Patients have less than one complete spontaneous bowel movement per week
4. Patients rely on laxatives to assist defecation for a long time
5. More than 20% the radio-paque markers localized in the colon after 72 hours based on colonic transit studies
6. Patients were refractory to conservative treatment for more than 1 year
7. Patients with a strong desire for surgery

Exclusion criteria

1. Pregnant or breast-feeding women
2. Patients with megacolon, megarectum,severe spastic constipation, severe rectocele, rectal prolapse (Oxford Grade IV or above)
3. Patients with colorectal neoplasms
4. Patients with small intestinal slow transit
5. Patients with constipation-predominant irritable bowel syndrome
6. Patients with inflammatory bowel disease
7. Patients with ileostomy
8. Patients with severe psychiatric disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2022-03-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Wexner Constipation Score | From the pre-operation to 36 months following surgery
  The Wexner Constipation Score will be recorded in terms of scores. Questions examine constipation in its clinical expressions. Each question is answered on a scale of 0 to 4. The scale ranges from 0 (best) to 30 (worst)

SECONDARY OUTCOMES:
Gastrointestinal Quality of Life Index | From the pre-operation to 36 months following surgery
  Gastrointestinal Quality of Life Index will be recorded in terms of scores. There are The four possible answers to every question, scored from 0 points (worst) to 4 points (best). The final sum ranges from 0(worst) to 144(best).
36-item short-form health survey | From the pre-operation to 36 months following surgery
  There are eight spheres in the SF-36 survey, including physical function, role physical, role emotional, physical pain, vitality, mental health, social function and general health. Results of each sphere will be recorded in terms of scores. Once the questionnaire was applied to the patients, a summary calculation and a linear transformation were performed to obtain a score within a scale from 0(worst) to 100(best).
The incidence of complications | From the pre-operation to 36 months following surgery
  Postoperative complications includes short-term and long-term complications, such as ileus, anastomotic leak, small intestinal obstruction, constipation recurrence and so on. Number of Participants with complications will be recorded.
The number of bowel movements per week | From the pre-operation to 36 months following surgery
  The number of bowel movements will be recorded in terms of times per week.
Wexner's incontinence score | From the pre-operation to 36 months following surgery
  The Wexner's incontinence score will be recorded in terms of scores. the sacles have 5 items to quantify incontinence grade and frequency and its effect on ordinary life. Each question is answered on a scale of 0 to 4, the global score ranging from 0 (best) to 20 (worst).
The incidence of abdominal pain | From the pre-operation to 36 months following surgery
  The incidence of abdominal pain will be recorded in terms of percent. no special measurement is needed.
The incidence of bloating | From the pre-operation to 36 months following surgery
  The incidence of bloating will be recorded in terms of percent
The incidence of diarrhea | From the pre-operation to 36 months following surgery
  The incidence of diarrhea will be recorded in terms of percent.
The incidence of straining | From the pre-operation to 36 months following surgery
  The incidence of straining will be recorded in terms of percent.
The incidence of laxative use | From the pre-operation to 36 months following surgery
  The incidence of laxative use will be recorded in terms of percent.
The incidence of enema use | From the pre-operation to 36 months following surgery
  The incidence of enema use use will be recorded in terms of percent.
Intraoperative measures | Perioperative period
  Operation time (minutes), blood loss (mL), complications (classified according to Clavien-Dindo) for both study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Tong, MD, Study Director — Army Medical Center (Daping Hospital)
Locations (16):
- China (16):
  - Army Medical Center (Daping Hospital), Yuzhong, Chongqing Municipality
  - No. 940 Hospital of Joint Logistics Support Force of Chinese People's Liberation Army, Lanzhou, Gansu
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - General Hospital of the Eastern Theater Cammand of the PLA, Nanjing, Jiangsu
  - The First Hospital of China Medical University, Shengyang, Liaoning
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Renji Hospital, Shanghai Jiaotong University, Pudong, Shanghai Municipality
  - Shanghai Pudong New Area People's Hospital, Pudong, Shanghai Municipality
  - Xijing Hospital, Xi’an, Shanxi
  - Chengdu Analrectal Hospital, Chengdu, Sichuan
  - The General Hospital of Western Theater Command, Chengdu, Sichuan
  - The Second People's Hospital of Yibin, Yibin, Sichuan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Macha MR. The feasibility of laparoscopic subtotal colectomy with cecorectal anastomosis in community practice for slow transit constipation. Am J Surg. 2019 May;217(5):974-978. doi: 10.1016/j.amjsurg.2019.03.018. Epub 2019 Mar 26. PMID 30948148
- [Result] Wei D, Cai J, Yang Y, Zhao T, Zhang H, Zhang C, Zhang Y, Zhang J, Cai F. A prospective comparison of short term results and functional recovery after laparoscopic subtotal colectomy and antiperistaltic cecorectal anastomosis with short colonic reservoir vs. long colonic reservoir. BMC Gastroenterol. 2015 Mar 18;15:30. doi: 10.1186/s12876-015-0257-7. PMID 25887580
- [Result] Perivoliotis K, Baloyiannis I, Tzovaras G. Cecorectal (CRA) versus ileorectal (IRA) anastomosis after colectomy for slow transit constipation (STC): a meta-analysis. Int J Colorectal Dis. 2022 Mar;37(3):531-539. doi: 10.1007/s00384-022-04093-y. Epub 2022 Jan 12. PMID 35020001
- [Result] Knowles CH, Grossi U, Horrocks EJ, Pares D, Vollebregt PF, Chapman M, Brown S, Mercer-Jones M, Williams AB, Yiannakou Y, Hooper RJ, Stevens N, Mason J; NIHR CapaCiTY working group; Pelvic floor Society and; European Society of Coloproctology. Surgery for constipation: systematic review and practice recommendations: Graded practice and future research recommendations. Colorectal Dis. 2017 Sep;19 Suppl 3:101-113. doi: 10.1111/codi.13775. PMID 28960922
- [Result] Deng XM, Zhu TY, Wang GJ, Gao BL, Li RX, Wang JT. Laparoscopic total colectomy with ileorectal anastomosis and subtotal colectomy with antiperistaltic cecorectal anastomosis for slow transit constipation. Updates Surg. 2023 Jun;75(4):871-880. doi: 10.1007/s13304-023-01458-y. Epub 2023 Mar 14. PMID 36914915
- [Derived] Tian Y, Guo M, Bu F, Ni L, Liu W, Gao F, Lan H, Cui Z, Fu T, Wang Y, Li F, Xu D, Gao H, Zhang L, Liu X, Huang B, Wang L, Jiang C, Jiang J, Gong W, Tong W. Total colectomy with ileorectal anastomosis versus subtotal colectomy with cecal-rectal anastomosis for slow transit constipation: protocol for a multicenter randomized controlled trial (STOPS trial). Trials. 2025 Oct 10;26(1):402. doi: 10.1186/s13063-025-09049-5. PMID 41074220